CLINICAL TRIAL: NCT04136535
Title: A Multicenter, Randomized, Phase II Study of Pemetrexed and Carboplatin With or Without Anlotinib Hydrochloride for Advanced or Locally-advanced Osimertinib-resistant Non-squamous Non-small Cell Lung Cancer (ALTER-L031)
Brief Title: Pemetrexed and Carboplatin With or Without Anlotinib Hydrochloride for Osimertinib-resistant Non-squamous NSCLC
Acronym: PCA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, primary care physician, Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L031
Record Dates: First submitted 2019-10-14; First posted 2019-10-23 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pemetrexed and Carboplatin with Anlotinib (Experimental): Pemetrexed and Carboplatin with Anlotinib
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Anlotinib
- Pemetrexed and Carboplatin without Anlotinib (Active Comparator): Pemetrexed and Carboplatin without Anlotinib
  Interventions: Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed，500mg/m²，ivgtt ，d1，q3w
Drug: Carboplatin — Carboplatin，AUC 5.0，ivgtt，d1，q3w，
Drug: Anlotinib — Anlotinib ，12 mg，po，qd，d1-14，q3w；
  Arms: Pemetrexed and Carboplatin with Anlotinib

SUMMARY:
Evaluate the efficacy and safety of Anlotinib Hydrochloride in combination with Pemetrexed and Carboplatin versus Pemetrexed and Carboplatin for advanced or locally-advanced Osimertinib-resistant non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
Anlotinib Hydrochloride in combination with Pemetrexed and Carboplatin use 4 cycles,then continue pem and anlotinib until PD

Pemetrexed and Carboplatin use 4 cycles,then continue pem until PD

TO see the different of PFS and OS and safety between the two group

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years to 75 Years patients voluntarily participate in this study, signed and dated informed consent with good compliance and follow-up; 2. Confirmed as locally advanced and / or metastatic non-squamous non-small cell lung cancer (NSCLC) by cytology or histology, the diagnosis should be completed at least 6 months after the end of chemotherapy if adjuvant chemotherapy and / or neoadjuvant chemotherapy received (diagnosis based on sputum smear is not accepted) ; 3. Presence of EGFR activating mutations and previously disease progression to Osimertinib (previously treated with 1st / 2nd generation EGFR-TKI or not)； 4. At least one target lesion that has accurate measurement by magnetic resonance imaging (MRI) or computed tomography (CT) (conventional CT≥20 mm or spiral CT≥10 mm) in at least 1 direction; 5. Life expectancy is at least 3 months; 6. ECOG PS Scoring: 0~1 point; 8. The main organs function are normally, the following criteria are met:

Blood routine examination criteria (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli):

i) hemoglobin (HB) ≥90g/L ii) neutrophil absolute (ANC) ≥1.5×109/L iii) platelet (PLT) ≥80×109/L Biochemical tests meet the following criteria i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; iii) serum creatinine (Cr) ≤1.25 ULN or creatinine clearance (CCr)≥45mL/min (Cockcroft-Gault formula).

9.Female patients of childbearing age agree that contraceptive measures must be used within the study period and within 8 weeks after the end of the study drug treatment. The serum or urine test indicates unpregnancy within 7 days prior to the study. Male patients agree to have contraceptive use during the study period and within 8 weeks after the end of the study period or have had surgical sterilization.

Exclusion Criteria:

1. Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer) and lung adenosquamous carcinoma mixed with squamous carcinoma;
2. Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 21 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms);
3. Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel and the distance between tumor and bronchial tree is ≤ 2 cm; or there is a significant pulmonary cavity or necrotizing tumor;
4. Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg after optimal medical treatment);
5. Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
6. Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
7. Urine routine test protein ≥++, and confirmed 24 hours urine protein> 1.0 g;
8. There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
9. Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
10. Long-term unhealed wounds or fractures;
11. Serious infection (≥CTC AE Level 2 infection) requiring systemic antibiotics;
12. decompensated diabetes or other ailments treated with high doses of glucocorticoids;
13. Active or chronic hepatitis C or/and hepatitis B infection;
14. Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
15. Patients have undergone major surgery within 4 weeks before enrollment or have severe trauma, fracture and ulcer;
16. Severe weight loss (greater than 10%) within 6 weeks prior to enrollment;
17. Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
18. Events of venous/ arterious thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
19. Patients have contraindication to platinum drugs (Cisplatin/Carboplatin) and cytotoxic drug (Pemetrexed);
20. Patients have anaphylactic reaction due to Anlotinib Hydrochloride or the excipient in investigational drug.
21. Planned for systemic anti-tumor therapy during the study period or within 4 weeks prior to enrollment, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or use mitomycin C within 6 weeks prior to receiving investigational drug). Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks before enrollment or limited-field radiotherapy was performed for planned tumor lesions within 2 weeks before enrollment.
22. Patients with other situations which are not suitable for the study according to the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  Progress free survival

CONTACTS AND LOCATIONS:
Overall Officials: chang j hua, PD, Principal Investigator — PI
Locations (1):
- Caner hospital & Shenzhen Hospital, Chinese Academy of Medical Sciences and Peking Uninon Medical college, Shenzhen, shenzhen, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700